CLINICAL TRIAL: NCT03330782
Title: Effect-site Concentration of Remifentanil for Preventing Propofol Injection Pain in Elderly Patients: A Comparison With Adult Patients
Brief Title: Remifentanil for Preventing Propofol Injection Pain in Elderly Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ajou University School of Medicine (Other)
Responsible Party: Principal Investigator, Jong Yeop Kim, Professor, Ajou University School of Medicine
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: AJIRB-MED-OBS-17-197
Record Dates: First submitted 2017-10-30; First posted 2017-11-06 (Actual); Last update posted 2019-07-05 (Actual); Status verified 2019-07

CONDITIONS: Drug Usage
Keywords: pain; propofol; remifentanil
MeSH Terms: conditions — Pain | interventions — Remifentanil

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Elderly (Experimental): Remifentanil was infused at predetermined effect-site concentration before propofol infusion in elderly patients.
  Interventions: Drug: Remifentanil
- Adult (Active Comparator): Remifentanil was infused at predetermined effect-site concentration before propofol infusion in adult patients.
  Interventions: Drug: Remifentanil

INTERVENTIONS:
Drug: Remifentanil — Remifentanil was infused at predetermined effect-site concentration prior to propofol infusion (initial concentration: 3.0 ng/ml) in elderly patients (65-80 years)
  Other Names: Ultiva
  Arms: Elderly
Drug: Remifentanil — Remifentanil was infused at predetermined effect-site concentration prior to propofol infusion (initial concentration: 3.0 ng/ml) in adult patients (20-60 years)
  Other Names: Ultiva
  Arms: Adult

SUMMARY:
Elderly patients show different pharmacokinetic and pharmacodynamic variables and usually need smaller doses of anesthetic drugs than younger patients. The purpose of this study was to investigate the optimal effect-site concentration of remifentanil for preventing injection pain during propofol induction in elderly patients by the Dixon's up-and-down method.

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status I or II undergoing general anesthesia

Exclusion Criteria:

* neurologic disorder
* psychologic disorder
* vascular disorder
* patients with chronic pain
* difficulty in vascular access

Ages: 19 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2017-11-16 (Actual); Primary Completion 2018-06-15 (Actual); Study Completion 2018-06-15 (Actual)

PRIMARY OUTCOMES:
Severity of propofol injection pain-4 point scale | during 3 min after remifentanil and propofol infusion to reach the equilibrium of plasma and effect-site concentration
  0 = no pain (negative response to questioning),
  1. = mild pain (pain reported only in response to questioning without any behavioral signs),
  2. = moderate pain (pain reported in response to questioning and accompanied by a behavioral signs or pain reported spontane¬ously without questioning),
  3. = severe pain (vocal response accompanied by facial grimacing, arm withdrawal, or tears)

CONTACTS AND LOCATIONS:
Overall Officials: Jong Yeop Kim, Principal Investigator — Ajou University Hospital, Suwon, Gyeongki-do, South Korea, 443-721
Locations (1):
- Jong Yeop Kim, Suwon, Gyeonggi-do, South Korea